CLINICAL TRIAL: NCT06617091
Title: A Phase 1 Randomized Double Blinded Placebo Controlled, Dose Ranging Trial, of a Gorilla Adenovirus Vectored Networked Epitopes Vaccine, Administered to Healthy Adults Living Without HIV and Living With HIV, in Southern Africa
Brief Title: A Trial of a Gorilla Adenovirus Vectored Networked Epitopes Vaccine, Administered to Healthy Adults Living Without and With HIV.
Acronym: IAVI C114
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Ragon Institute (Unknown); ReiThera Srl (Industry); Mutala Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IAVI C114
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: HIV
Keywords: GRAdHIVNE1 Vaccine
MeSH Terms: interventions — Disease Vectors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized controlled Double - blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People living with HIV (PLWH) and People living without HIV (PLWoH) (Experimental): Participants living without HIV (PLWoH) will be assigned to receive either a single dose, 2 doses of the GRAdHIVNE1 vaccine, or placebo. Participants living with HIV (PLWH) will be assigned to receive either 2 doses of the GRAdHIVNE1 vaccine, or placebo.
  Each participant is to receive GRAdHIVNE1 at vaccine dose 5x10^10 or 2x10^11 or to receive placebo.
  Interventions: Drug: GRAdHIVNE1 Vaccine
- Placebo NaCl for injection (Placebo Comparator): Participants living without HIV (PLWoH) will be assigned to receive either a single dose, 2 doses of the GRAdHIVNE1 vaccine, or placebo. Participants living with HIV (PLWH) will be assigned to receive either 2 doses of the GRAdHIVNE1 vaccine, or placebo.
  Each participant is to receive GRAdHIVNE1 at vaccine dose 5x10^10 or 2x10^11 or to receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GRAdHIVNE1 Vaccine — This is a dose ranging study that will allow for simultaneous enrollment of participants in both low and high dose groups.
  Other Names: gorilla-isolated adenovirus (GRAd32) vector
  Arms: People living with HIV (PLWH) and People living without HIV (PLWoH)
Other: Placebo — This is a dose ranging study that will allow for simultaneous enrollment of participants in both low and high dose groups.
  Arms: Placebo NaCl for injection

SUMMARY:
A Phase 1 Randomized Double Blinded Placebo Controlled, Dose Ranging Trial, of a Gorilla Adenovirus Vectored Networked Epitopes Vaccine (GRAdHIVNE1 Vaccine), Administered to Healthy Adults Living without HIV and Living with HIV, in Southern Africa

DETAILED DESCRIPTION:
This is a Phase 1 trial for the GRAdHIVNE1 vaccine, designed to evaluate safety, tolerability, and immunogenicity in healthy individuals (PLWoH) including healthy People Living with HIV (PLWH). This study builds on insights from prior T-cell vaccine trials and pre-clinical non-human primate studies, which demonstrated that robust CD8+ T cell responses, are crucial for viral control but require broad, polyfunctional responses that can also effectively counteract HIV's diversity and immune evasion strategies. Inclusion of PLWoH and PLWH in this study is important for safety, tolerability and immunogenicity data that can inform further development of the vaccine for prevention and therapeutic use. Prior clinical trials, using adenovirus vectors and exploring different vaccine approaches, demonstrated safety and potential immunogenic benefits in PLWH, despite not achieving sustained viral suppression post-treatment interruption Understanding these dynamics is key to evaluating the full therapeutic potential of vaccine induced immune responses in controlling HIV as well as inform the potential of the vaccine in aborting the establishment of a disseminated infection in the setting of prevention.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age on the day of screening and has not reached his or her 51st birthday on the day of signing the Informed Consent Document.
2. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
3. In the opinion of the Principal Investigator or designee and based on Assessment of Informed Consent Understanding results, has understood the information provided and potential impact and/or risks linked to administration of the investigational product; written informed consent will be obtained from the participant before any study-related procedures are performed.
4. All sexually active female participants capable of becoming pregnant must commit to use an effective method of contraception from 21 days prior to receiving the IP until 4 months following the last IP administration, including:

   1. Intrauterine device, or contraceptive implant
   2. Hormonal contraception
   3. Successful vasectomy in the male partner (considered successful if a woman reports that a male partner has [1] documentation of azoospermia by microscopy (< 1 year ago), or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post-vasectomy)
5. Women who have undergone a hysterectomy, bilateral oophorectomy, or tubal ligation, as well as those who are postmenopausal (> 45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone [FSH] level > 40 IU/L) will not be required to use contraceptives.
6. Willing to forgo donations of blood, or any other tissues during the study.

   Additional Inclusion criteria for PLWH
7. Confirmed HIV infection (HIV Ab+ or HIV RNA+) by documentation in the medical records or in-clinic HIV testing on screening visit.
8. CD4 ≥ 500 cells/µl at screening.
9. Currently on ART, and documentation of continuous combination ART (cART) for at least 12 months with suppression of plasma HIV-1 viral load < 50 copies / ml for greater than 6 months prior to trial entry, measured on at least 2 independent occasions that can include the screening viral load. cART is defined as a regimen including ≥ 2 compounds, e.g., 2 nucleoside reverse transcriptase inhibitors plus either non-nucleoside reverse transcriptase inhibitor or protease inhibitor or integrase inhibitor.
10. Viral load < 50 copies / ml at time of screening (within 28 days prior to IP administration).
11. Must commit to adhering to a suppressive ART regimen for the duration of the study

Exclusion Criteria:

1. Any clinically significant acute or chronic medical condition, other than HIV infection (in Part B only), that is considered progressive or in the opinion of the investigator makes the participant unsuitable for participation in the study.
2. For the PLWH (Part B), history of AIDS-defining illness or CD4 < 200 cells/µl.
3. If female, pregnant, lactating or planning a pregnancy during the period of screening through completion of the study.
4. In the past 6 months a history of alcohol or substance use, judged by the Investigator to potentially interfere with participant study compliance.

Bleeding disorder that was diagnosed by a physician (e.g., Factor deficiency, coagulopathy or platelet disorder that requires special precautions). Note: A participant who states that he or she has easy bruising or bleeding but does not have a formal diagnosis and has intramuscular injections and blood draws without any adverse experience, is eligible.

6. History of a splenectomy. 7. Previous receipt of an adenovirus vectored vaccine. 8. Receipt of live attenuated vaccine or other vaccine within the previous 60 days or planned receipt within 180 days after administration of IP. Receipt of blood transfusion or blood derived products within the previous 3 months.

9. Participation in another clinical trial of an investigational product currently, within the previous 3 months or expected participation during this study.

10. Prior receipt of an investigational HIV vaccine candidate, monoclonal antibody or polyclonal immunoglobulin (note: receipt of placebo in a previous HIV vaccine or monoclonal antibody trial will not exclude a participant from participation if documentation is available and the Medical Monitor gives approval).

11. History of severe local or systemic reactogenicity to vaccines (e.g., anaphylaxis, respiratory difficulties, angioedema).

12. Psychiatric condition that compromises safety of the participant and precludes compliance with the protocol. Specifically excluded are persons with history of psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.

13. If, in the opinion of the Principal Investigator or designee, it is not in the best interest of the participant to participate in the trial.

14. Seizure disorder: a participant who has had a seizure in the last 3 years is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for 3 years.) 15. Infectious disease: chronic hepatitis B infection (HbsAg positive), current hepatitis C infection (HCV Ab positive and/ or HCV RNA) or treatment for hepatitis C infection in the past year, or active syphilis (RPR confirmed by TPHA).

16. A history of malignancy within the past 5 years (prior to screening) or ongoing malignancy.

17. Active, serious infections (other than HIV infection in PLWH) requiring parenteral antibiotic, antiviral or antifungal therapy within 30 days prior to enrollment.

18. Any abnormal laboratory parameters at screening per protocol. 19. Any clinically relevant abnormality on history or examination including history of immunodeficiency or autoimmune disease, other than HIV among the PLWH; use of systemic corticosteroids, immunosuppressive, anticancer, or other medications considered significant by the investigator within the previous 6 months.

Eligibility Criteria Specific to PLWoH (Part A) People living without HIV(PLWoH) at screening, must be deemed to be at low risk of HIV infection and willing to maintain low-risk behavior for the duration of the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Assess safety and tolerability of GRAdHIVNE1 vaccine | 7 Day
  1. Proportion of participants with each type of reactogenicity event classified by severity of the events from initial administration through 7 days following completion of each dose of the investigational product.
Assessment of unsolicited adverse events (AEs) | 28 day
  Proportion of participants reporting unsolicited adverse events (AEs), including safety laboratory (biochemical, hematological) parameters, classified by severity and causality, from initial administration through 28 days following completion of each dose of the investigational product.
Assessment of SAEs | 19 months
  Proportion of participants reporting serious adverse events (SAEs) throughout the study period, classified by causality.

SECONDARY OUTCOMES:
To evaluate cellular immune responses elicited by GRAdHIVNE1 vaccine. | 19 Months
  1. Response rate and magnitude of the vaccine induced HIV specific T cell response at peak immunogenicity as measured by intracellular cytokine staining assay or IFNγ ELISpot assay after each dose.
To evaluate cellular immune responses elicited by GRAdHIVNE1 vaccine. | 19 months
  To assess antigen specific proliferative memory T cell responses induced by vaccination.
To evaluate cellular immune responses elicited by GRAdHIVNE1 vaccine. | 19 months
  To identify immunogenic epitopes within the vaccine immunogen and define the HLA restriction.
To evaluate cellular immune responses elicited by GRAdHIVNE1 vaccine. | 19 months
  To define the functional characteristics of antigen specific T cells by assessing proliferation, cytotoxicity, tetramer analysis and TCR sequences.
To evaluate cellular immune responses elicited by GRAdHIVNE1 vaccine. | 19 months
  To evaluate vaccine induced innate immune responses.
To evaluate cellular immune responses elicited by GRAdHIVNE1 vaccine. | 19 months
  To characterize vaccine induced de novo T-cell responses compared to pre-existing responses in PLWH (Part B).
To evaluate cellular immune responses elicited by GRAdHIVNE1 vaccine. | 19 months
  To conduct analyses to further understand HIV and vaccine immunology

CONTACTS AND LOCATIONS:
Overall Officials: Theodorah Ndzhukule, Principal Investigator — Desmond Tutu Health Foundation; Limakatso Lebina, Principal Investigator — Africa Health Research Institute (AHRI); Tariro Makadzange, Principal Investigator — Mutala Trust
Locations (3):
- South Africa (2):
  - AHRI, Mtubatuba, KwaZulu-Natal
  - DTHF, Cape Town, Western Cape
- Mutala, Harare, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
The full data package will be made available to the public approximately 12 months after the trial Completion.
  To protect participant privacy the data package will be sent to a company who specializes in anonymization and pseudonymization of clinical trial data that will strip out or anonymize any potential identifying information such as participant IDs, dates of birth, initials, visit dates, or any other data that alone or in aggregate could identify an individual.
Supporting Information: Study Protocol
Time Frame: Once the final anonymized data package is available it will be posted to the Vivli data repository platform. Vivli will make data available for researchers for 7 years, unless they are contractually unable to do so.
Access Criteria: Vivli utilizes an independent peer review process to evaluate the validity of external requests. Criteria include the intended analysis by the requestors, professional credentials of the requestors, and the feasibility of the proposed work based on the data requested. After approval by the peer review board, the requestors must sign a data transfer agreement before the data are provided. The data transfer agreement will require the requestor to specify how the transferred data will be held in secure, controlled access during the analysis interval.